CLINICAL TRIAL: NCT00000832
Title: A Randomized, Placebo-Controlled, Double-Blinded Phase I Safety and Immunogenicity Trial of Recombinant Envelope Protein, HIV-1 SF-2 rgp120 (BIOCINE), Combined With MF59 in HIV-1 Uninfected Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Prevention
Other Study IDs: AVEG 024; 10575 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; HIV-1; Adjuvants, Immunologic; HIV Envelope Protein gp120; AIDS Vaccines; HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections | interventions — MF59 oil emulsion

INTERVENTIONS:
Biological: MF59
Biological: rgp120/HIV-1 SF-2

SUMMARY:
To determine the safety and immunogenicity of rgp120/HIV-1SF2 combined with MF59 adjuvant emulsion versus MF59 alone in HIV-negative volunteers.

One approach to improve the immunogenicity of an HIV-1 subunit protein vaccine is to combine the immunogen with an adjuvant.

DETAILED DESCRIPTION:
One approach to improve the immunogenicity of an HIV-1 subunit protein vaccine is to combine the immunogen with an adjuvant.

Healthy volunteers receive intramuscular injections of rgp120/HIV-1SF2 with MF59 adjuvant emulsion or MF59 alone at months 0, 1, 6, 9, 10 and 12 (was months 0, 1, 6 and 10, amended 12/19/96).

ELIGIBILITY:
Inclusion Criteria

Volunteers must have:

* Normal history and physical exam.
* HIV negativity.
* Absolute CD4 count >= 400 cells/mm3.
* Normal urine dipstick with esterase and nitrite.
* Lower risk sexual behavior.

Exclusion Criteria

Co-existing Condition:

Subjects with the following symptoms or conditions are excluded:

* Positive hepatitis B surface antigen.
* Medical or psychiatric condition (such as recent suicidal ideation or present psychosis) that precludes compliance.
* Active syphilis. NOTE: Subjects with serology documented to be a false positive or due to a remote (> 6 months) treated infection are eligible.
* Active tuberculosis. NOTE: Subjects with a positive PPD and a normal chest x-ray showing no evidence of TB and not requiring isoniazid therapy are eligible.

Subjects with the following prior conditions are excluded:

* History of immunodeficiency, chronic illness, autoimmune disease, or use of immunosuppressive medications.
* History of anaphylaxis or other serious adverse reactions to vaccines.
* History of serious allergic reaction to any substance, requiring hospitalization or emergent medical care (e.g., Stevens-Johnson syndrome, bronchospasm, or hypotension).
* Prior psychiatric condition (such as history of suicide attempts or past psychosis) that precludes compliance.
* History of cancer unless there has been surgical excision that is considered to have achieved cure.

Prior Medication:

Excluded:

* Live attenuated vaccines within 60 days prior to study entry. NOTE: Medically indicated killed or subunit vaccines (e.g., influenza, pneumococcal) do not exclude if administered at least 2 weeks from HIV immunizations.
* Experimental agents within 30 days prior to study entry.
* Prior HIV vaccines.

Prior Treatment:

Excluded:

* Blood products or immunoglobulin within the past 6 months.

Identifiable high-risk behavior for HIV infection, including:

* History of injection drug use within past 12 months.
* Higher risk sexual behavior.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Study Completion 1998-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corey L, Study Chair
Locations (4):
- United States (4):
  - UAB AVEG, Birmingham, Alabama
  - St. Louis Univ. School of Medicine AVEG, St Louis, Missouri
  - Univ. of Rochester AVEG, Rochester, New York
  - JHU AVEG, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Corey L, Weinhold K, Montefiori D, Stablein D. CTL and neutralizing antibody responses with a combination HIV-1 vaccine regimen. Int Conf AIDS. 1998;12:636 (abstract no 33221)
- [Background] Kahn JO, Sinangil F, Baenziger J, Murcar N, Wynne D, Coleman RL, Steimer KS, Dekker CL, Chernoff D. Clinical and immunologic responses to human immunodeficiency virus (HIV) type 1SF2 gp120 subunit vaccine combined with MF59 adjuvant with or without muramyl tripeptide dipalmitoyl phosphatidylethanolamine in non-HIV-infected human volunteers. J Infect Dis. 1994 Nov;170(5):1288-91. doi: 10.1093/infdis/170.5.1288. PMID 7963729